CLINICAL TRIAL: NCT07240454
Title: Safety and Efficacy of Aspirin Continuation or Discontinuation in Conservative Treatment for Chronic Subdural Hematoma: A Randomized Clinical Trial
Brief Title: Aspirin Continuation or Discontinuation in Conservative Treatment for Chronic Subdural Hematoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tao Liu (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Tao Liu, MD, The George Institute
Organization: The George Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aspirin CSDH
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; Aspirin; Conservative Treatment; Randomized Clinical Trial; Safety; Efficacy; cSDH
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin Continuation Group (Experimental): All participants received standard conservative treatment for chronic subdural hematoma, with a randomized intervention to continue aspirin administration. This group of participants received oral administration of aspirin at a dose of 100 mg per day.
  Interventions: Drug: Aspirin Continuation
- Aspirin Discontinuation Group (Experimental): All participants received standard conservative treatment for chronic subdural hematoma, with a randomized intervention to discontinue aspirin administration. This group of participants did not use aspirin during the treatment period.
  Interventions: Drug: Aspirin Discontinuation

INTERVENTIONS:
Drug: Aspirin Continuation — All participants received standard conservative treatment for chronic subdural hematoma, with a randomized intervention to continue aspirin administration. This group of participants received oral administration of aspirin at a dose of 100 mg per day.
  Arms: Aspirin Continuation Group
Drug: Aspirin Discontinuation — All participants received standard conservative treatment for chronic subdural hematoma, with a randomized intervention to discontinue aspirin administration. This group of participants did not use aspirin during the treatment period.
  Arms: Aspirin Discontinuation Group

SUMMARY:
This clinical study aims to learn about the efficacy and safety of aspirin continuation or discontinuation in conservative treatment for chronic subdural hematoma. All participants received standard conservative treatment for chronic subdural hematoma, with a randomized intervention to either continue or discontinue aspirin administration. By participating in this study, participants can receive additional scientific guidance on aspirin medication management beyond routine conservative treatment, thereby optimizing individualized therapy.

DETAILED DESCRIPTION:
Chronic subdural hematoma is a common condition in neurosurgery, predominantly affecting the elderly. Its incidence increases with age, often developing gradually following minor head trauma. Clinical manifestations vary widely, with severe cases potentially leading to coma or even death, imposing a significant burden on patients and their families.

Current treatment approaches for chronic subdural hematoma include surgical intervention and conservative management. Conservative treatment is suitable for some patients with milder conditions or high surgical risk, primarily involving bed rest and medication. However, its efficacy varies among individuals, and close monitoring for multiple potential complications is essential throughout the treatment process.

Aspirin, a commonly used antiplatelet agent, is widely applied in the prevention and treatment of cardiovascular and cerebrovascular diseases. Its use in chronic subdural hematoma patients presents complexities: some patients had been taking aspirin long-term prior to onset. Whether to continue aspirin during conservative management remains controversial, necessitating further research to clarify its safety and efficacy. Continuing the medication may increase the risk of hematoma enlargement, while discontinuation may trigger thromboembolic events.

For cSDH patients on long-term aspirin therapy who opt for conservative management, there is currently no guideline or consensus on "continue vs. discontinue." Clinical decisions are often made by multidisciplinary teams (MDTs) based on individualized risk assessment of bleeding versus thrombosis (with a higher rate of discontinuation strategies). A randomized controlled trial in surgical patients (JAMA Neurology, 2025) showed that discontinuing aspirin after surgery did not reduce 6-month recurrence, and discontinuation-related complications showed no significant difference, suggesting that a "one-size-fits-all" discontinuation approach is unreasonable. However, this evidence cannot be extrapolated to the conservative treatment population, making the conduct of this RCT practically necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female;
* Confirmed diagnosis of chronic subdural hematoma (cSDH) by cranial CT and/or MRI;
* Intended for conservative management (i.e., no surgical evacuation indication at enrollment);
* Regular aspirin use at enrollment;
* Informed consent signed by the patient or legal representative.

Exclusion Criteria:

* Patients requiring emergency surgery to remove hematoma at enrollment;
* Concurrent use of other anticoagulants or antiplatelet agents that cannot be discontinued according to the study protocol;
* cSDH secondary to other diseases or conditions (e.g., excessive drainage from ventriculoperitoneal shunts, intracranial tumors);
* Active bleeding events or major cardiac events (e.g., acute myocardial infarction, unstable angina, or revascularization surgery) within 30 days prior to enrollment;
* Known bleeding disorders (e.g., hemophilia, severe thrombocytopenia);
* Individuals unable to provide informed consent or for whom completion of follow-up is anticipated to be difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
recurrence or progression of the subdural hematoma | 6 months
  The primary outcome was defined as recurrence or progression of the subdural hematoma at 6 months, confirmed by positive radiological findings with or without associated clinical symptoms, necessitating additional pharmacological or surgical intervention. Positive radiological findings were defined as reappearance of ipsilateral CSDH with a midline shift greater than 5 mm at 6 months；a maximum hematoma thickness exceeding 10 mm at 6 months; or an increase in maximum hematoma thickness of more than 3 mm.

SECONDARY OUTCOMES:
modified Rankin Score (mRS) | at 6 months
  0=no symptoms, 1=no significant disability, 2=slight disability, 3= moderate disability, 4=moderate severe disability, 5=severe disability, 6=death
Surgical conversion rate | at 6 months
mortality | at 6 months
Peripheral vascular events | 6 months
  Peripheral vascular events: including peripheral arterial occlusion (PAO), thromboembolic events (deep vein thrombosis, pulmonary embolism), and other peripheral hemorrhagic events.
Acute cardiovascular and cerebrovascular events | 6 months
  Acute cardiovascular and cerebrovascular events: including stroke (hemorrhagic stroke, ischemic stroke), or cardiovascular events such as myocardial infarction or injury (PMI), ST-segment elevation myocardial injury (STEMI), and non-ST-segment elevation myocardial infarction (NSTEMI).
new-onset contralateral chronic subdural hematoma | 6 months
Change in hematoma volume | 6 months
EQ-5D-5L Questionnaire | 6 months
  EuroQol Group 5-Dimension 5-Level Self-Report Questionnaire
Montreal Cognitive Assessment Scale | 6 months
  Use the MoCA scale to assess cognitive function.
Red Blood Cell Lifespan | 6 months
Other adverse events | 6 months
  Other adverse events: including liver and kidney function abnormalities, infections, anemia, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided